CLINICAL TRIAL: NCT07253519
Title: The Relationship Between Mood and Insomnia Severity and Caregiver Burden in Caregivers of Stroke Patients
Brief Title: The Relationship Between Mood and Insomnia Severity and Caregiver Burden in Caregivers of Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: istftrrrr
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study will include stroke patients aged 18-80 years and their caregivers. Demographic data such as age, height, weight, and comorbidities will be recorded, along with stroke-specific characteristics including duration of stroke, affected side, lesion location, and etiology. Patients' functional status will be assessed using the Modified Rankin Scale, Brunnstrom Stages, and the Modified Barthel Index, while ambulation status will be documented with the Holden Scale. Caregivers will complete the Insomnia Severity Index to assess the severity of sleep disturbances and the Hospital Anxiety and Depression Scale to evaluate anxiety and depressive symptoms. Caregiver burden will be measured using the Zarit Caregiver Burden Scale. The study aims to investigate the relationship between caregivers' mood, insomnia severity, and caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Clinical diagnosis of stroke (ischemic or hemorrhagic; first-ever or recurrent).
* Ability of both the patient and caregiver to communicate in Turkish and participate in evaluations (mRS, Brunnstrom, Modified Barthel Index, Holden).
* Caregiver must have been the primary caregiver for the patient for at least 1 month.
* Willingness of both the patient and caregiver to participate in the study.

Exclusion Criteria:

* History of subarachnoid hemorrhage.
* Inability to communicate effectively due to severe aphasia or severe cognitive impairment.
* Terminal illness (life expectancy < 6 months).
* Inability to reliably complete questionnaires due to a psychiatric disorder.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stroke
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Zarit Caregiver Burden Scale (ZCBS) | Baseline
  Measures the perceived caregiver burden related to physical, emotional, social, and financial strain.
  Score Range: 0-88
  Higher scores indicate higher caregiver burden.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline
  Assesses the severity of insomnia symptoms experienced by caregivers. Score Range: 0-28
  Higher scores indicate more severe insomnia.
Hospital Anxiety and Depression Scale - Anxiety Subscale (HADS-A) | Baseline
  Evaluates the presence and severity of anxiety symptoms in caregivers. Score Range: 0-21
  Higher scores indicate more severe anxiety.
Hospital Anxiety and Depression Scale - Depression Subscale (HADS-D) | Baseline
  Assesses depressive symptom severity in caregivers. Score Range: 0-21
  Higher scores indicate more severe depression.
Modified Rankin Scale (mRS) | Baseline
  Clinician-rated scale assessing global disability in stroke patients. Score Range: 0-6
  Higher scores indicate greater disability.
Modified Barthel Index (MBI) | Baseline
  Measures independence in activities of daily living. Score Range: 0-100
  Higher scores indicate greater independence.
Holden Functional Ambulation Classification (FAC) | Baseline
  Evaluates ambulation ability and level of assistance required. Score Range: 0-5
  Higher scores indicate more independent walking.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)